CLINICAL TRIAL: NCT01745120
Title: A Phase 1/2 Open Label Study Evaluating the Safety and Efficacy of Gene Therapy in Subjects With β-Thalassemia Major by Transplantation of Autologous CD34+ Cells Transduced Ex Vivo With a Lentiviral βA-T87Q-Globin Vector (LentiGlobin® BB305 Drug Product)
Brief Title: A Study Evaluating the Safety and Efficacy of the LentiGlobin BB305 Drug Product in β-Thalassemia Major Participants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGB-204
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: β-thalassemia Major
Keywords: gene therapy; β thalassemia; hemoglobin; anemia; CD34
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LentiGlobin BB305 Drug Product (Experimental)
  Interventions: Genetic: LentiGlobin BB305 Drug Product

INTERVENTIONS:
Genetic: LentiGlobin BB305 Drug Product — Transplant of autologous hematopoietic stem cells transduced with LentiGlobin BB305 lentiviral vector.

SUMMARY:
This is a non-randomized, open label, multi-site, single-dose, phase 1/2 study in up to 18 participants (including at least 3 adolescents between 12 and 17 years of age, inclusive) with β-thalassemia major. The study will evaluate the safety and efficacy of autologous hematopoietic stem cell transplantation (HSCT) using LentiGlobin BB305 Drug Product [autologous CD34+ hematopoietic stem cells transduced with LentiGlobin BB305 lentiviral vector encoding the human βA-T87Q-globin gene].

DETAILED DESCRIPTION:
Subject participation for this study will be 2 years. Subjects who enroll in this study will be asked to participate in a subsequent long-term follow up study that will monitor the safety and efficacy of the treatment they receive for up to 13 years post-transplant.

ELIGIBILITY:
Inclusion criteria:

* Participants between 12 and 35 years of age, inclusive, at the time of consent/assent, and able to provide written consent/assent, if applicable.
* Diagnosis of β-thalassemia major and a history of at least 100 mL/kg/year of pRBCs or ≥8 transfusions of pRBCs per year for the prior 2 years.
* Eligible for allogeneic bone marrow transplant.
* Treated and followed for at least the past 2 years in a specialized center that maintained detailed medical records, including transfusion history.

Exclusion criteria:

* Positive for presence of human immunodeficiency virus type 1 or 2 (HIV 1 and HIV 2).
* A white blood cell (WBC) count <3 × 10^9/L, and / or platelet count <100 × 10^9/L if not due to hypersplenism.
* Uncorrected bleeding disorder.
* Any prior or current malignancy or myeloproliferative or immunodeficiency disorder.
* Immediate family member with a known or suspected Familial Cancer Syndrome (including but not limited to hereditary breast and ovarian cancer syndrome, hereditary non-polyposis colorectal cancer syndrome and familial adenomatous polyposis).
* Receipt of an allogeneic transplant.
* Advanced liver disease, including persistent aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin value >3 × the upper limit of normal, liver biopsy demonstrating cirrhosis, extensive bridging fibrosis, or active hepatitis.
* Kidney disease with a calculated creatinine clearance <30% normal value.
* Uncontrolled seizure disorder.
* Diffusion capacity of carbon monoxide (DLco) <50% of predicted (corrected for hemoglobin).
* A cardiac T2* <10 ms by magnetic resonance imaging (MRI).
* Any other evidence of severe iron overload that, in the Investigator's opinion, warrants exclusion.
* Clinically significant pulmonary hypertension, as defined by the requirement for ongoing pharmacologic treatment or the consistent or intermittent use of supplemental home oxygen.
* Participation in another clinical study with an investigational drug within 30 days of Screening.
* Any prior or current malignancy or myeloproliferative disorder.
* Prior receipt of gene therapy.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2013-08; Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Asmal, MD, Study Director — Genetix Biotherapeutics Inc.
Locations (6):
- United States (4):
  - Los Angeles, California
  - Oakland, California
  - Chicago, Illinois
  - Philadelphia, Pennsylvania
- Sydney, Australia
- Bangkok, Thailand

REFERENCES:
- [Derived] Thompson AA, Walters MC, Kwiatkowski J, Rasko JEJ, Ribeil JA, Hongeng S, Magrin E, Schiller GJ, Payen E, Semeraro M, Moshous D, Lefrere F, Puy H, Bourget P, Magnani A, Caccavelli L, Diana JS, Suarez F, Monpoux F, Brousse V, Poirot C, Brouzes C, Meritet JF, Pondarre C, Beuzard Y, Chretien S, Lefebvre T, Teachey DT, Anurathapan U, Ho PJ, von Kalle C, Kletzel M, Vichinsky E, Soni S, Veres G, Negre O, Ross RW, Davidson D, Petrusich A, Sandler L, Asmal M, Hermine O, De Montalembert M, Hacein-Bey-Abina S, Blanche S, Leboulch P, Cavazzana M. Gene Therapy in Patients with Transfusion-Dependent beta-Thalassemia. N Engl J Med. 2018 Apr 19;378(16):1479-1493. doi: 10.1056/NEJMoa1705342. PMID 29669226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in the United States, Australia and Thailand between 05 September 2013 (first participant first visit) and 21 February 2018 (last participant last visit).
Pre-assignment Details: A total of 19 participants were enrolled in the study and made up the Intent-to-Treat (ITT) population, which included all participants who initiated any study procedures, beginning with mobilization by granulocyte-colony stimulating factor (G-CSF), with or without plerixafor.
Groups:
- Non-β0/β0: Participants who had at least 1 mutation in the HBB gene that results in reduced but detectable expression of beta(β)-globin: β+ or βE (non-β0/β0 genotype) underwent hematopoietic stem cell (HSC) mobilization with G-CSF and plerixafor, followed by myeloablative conditioning and infusion with LentiGlobin BB305 Drug Product at a dose of greater than or equal to (>=) 3.0 × 10^6 CD34+ cells per kilogram (cells/kg).
- β0/β0: Participants who were bi-allelic for mutations in the HBB gene that results in absence of expression of β-globin: β0 (β0/β0 genotype) underwent HSC mobilization with G-CSF and plerixafor, followed by myeloablative conditioning and infusion with LentiGlobin BB305 Drug Product at a dose of >= 3.0 × 10^6 CD34+ cells/kg.
Period: Overall Study
Arm/Group | Non-β0/β0 | β0/β0
Started (Started = ITT) | 11 | 8
Completed | 10 | 8
Not Completed | 1 | 0
Not completed — Investigator decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (ITT) included all participants who initiated any study procedures, beginning with mobilization by G-CSF with or without plerixafor.
Groups:
- Non-β0/β0: Participants who had at least 1 mutation in the HBB gene that results in reduced but detectable expression of β-globin: β+ or βE (non-β0/β0 genotype) underwent HSC mobilization with G-CSF and plerixafor, followed by myeloablative conditioning and infusion with LentiGlobin BB305 Drug Product at a dose of >= 3.0 × 10^6 CD34+ cells/kg.
- Total: Total of all reporting groups
Arm/Group | Non-β0/β0 | β0/β0 | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of informed consent or assent (applicable for participants less than 18 years old) was reported
  Years | 22.7 (6.50) | 24.1 (7.62) | 23.3 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race of the participants was reported.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 8 | 6 | 14
    Black or African American | 0 | 0 | 0
    White | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Asian/Italian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Production of >=2.0 Grams Per Deciliter (g/dL) of Hemoglobin A (HbA) Containing βA-T87Q-globin (HbAT87Q) for the Six Months Between Month 18 and Month 24
Description: Percentage of participants with sustained production of >=2.0 grams per deciliter (g/dL) of hemoglobin A (HbA) containing βA-T87Q-globin (HbAT87Q) for 6 months (Month 18 to Month 24) was reported.
Time Frame: Month 18 to Month 24
Population: Transplant Population (TP) included all participants in the ITT population (participants who initiated any study procedures, beginning with mobilization by G-CSF with or without plerixafor) who underwent LentiGlobin BB305 Drug Product infusion.
Measure: Number; unit: Percentage of participants
Groups:
- Overall: Participants with a β0/β0 genotype or non-β0/β0 genotypes underwent HSC mobilization with G-CSF and plerixafor, followed by myeloablative conditioning and infusion with LentiGlobin BB305 Drug Product at a dose of >= 3.0 × 10^6 CD34+ cells/kg.
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Percentage of participants | 90.0 | 87.5 | 88.9

2. Primary Outcome: Percentage of Participants Who Achieved Transfusion Independence (TI)
Description: TI was defined as a weighted average hemoglobin (Hb) >= 9 g/dL without any packed red blood cells (pRBC) transfusions for a continuous period of >=12 months at any time during the study after LentiGlobin BB305 Drug Product infusion. Percentage of participants who achieved TI from time of drug product infusion up to 24 months was reported.
Time Frame: From time of drug product infusion up to 24 months
Population: TP included all participants in the ITT population (participants who initiated any study procedures, beginning with mobilization by G-CSF with or without plerixafor) who underwent LentiGlobin BB305 Drug Product infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Percentage of participants | 80.0 | 12.5 | 50.0

3. Secondary Outcome: Percentage of Participants Who Achieved Transfusion Independence (TI) at Month 18 and Month 24
Description: TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after LentiGlobin BB305 Drug Product infusion.
Time Frame: Month 18, Month 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Percentage of participants
  Month 18 | 80.0 | 12.5 | 50.0
  Month 24 | 80.0 | 0 | 44.4

4. Secondary Outcome: Duration of Transfusion Independence (TI)
Description: TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after LentiGlobin BB305 Drug Product infusion. Time period of TI will start when participants achieve a Hb >= 9 g/dL with no transfusions in the preceding 60 days. Duration of TI was calculated as the time from the start of TI (i.e. first Hb >= 9 g/dL with no transfusions in the preceding 60 days) up to the last available Hb at which the TI criteria are still met.
Time Frame: From time of drug product infusion up to 24 months
Population: TP included all participants in the ITT population (participants who initiated any study procedures, beginning with mobilization by G-CSF with or without plerixafor) who underwent LentiGlobin BB305 Drug Product infusion. Here, "number of participants analyzed" refers to the number of participants who reported TI.
Measure: Median (Full Range); unit: Months
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 8 | 1 | 9
Months | 18.91 [15.2 to 21.4] | 16.13 [16.13 to 16.13] | 17.28 [15.2 to 21.4]

5. Secondary Outcome: Time From LentiGlobin BB305 Drug Product Infusion to Last pRBC Transfusion Prior to Achieving Transfusion Independence (TI)
Description: TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after LentiGlobin BB305 Drug Product infusion. Time From LentiGlobin BB305 Drug Product Infusion to last pRBC transfusion prior to achieving TI was reported.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 8 | 1 | 9
Months | 2.00 [0.3 to 5.8] | 1.81 [1.81 to 1.81] | 1.81 [0.3 to 5.8]

6. Secondary Outcome: Time From LentiGlobin BB305 Drug Product Infusion to Achieving Transfusion Independence (TI)
Description: TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after LentiGlobin BB305 Drug Product infusion. Time from drug product infusion to initial achievement of TI was calculated as the time from drug product infusion to the first Hb at which a participant can be declared as TI.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 8 | 1 | 9
Months | 17.12 [15.0 to 20.9] | 17.51 [17.51 to 17.51] | 17.51 [15.0 to 20.9]

7. Secondary Outcome: Weighted Average Hemoglobin (Hb) During Period of Transfusion Independence (TI)
Description: The weighted average Hb is an average area under the curve during the period of TI, from the start of TI when the Hb is first >= 9 g/dL with no transfusions in the preceding 60 days to the last available Hb at which the TI criteria are still met. TI was defined as a weighted average Hb >= 9 g/dL without any pRBC transfusions for a continuous period of >= 12 months at any time during the study after LentiGlobin BB305 Drug Product infusion. Weighted average Hb during the period of TI was reported.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 8 | 1 | 9
Grams per deciliter (g/dL) | 10.44 (1.277) | 10.11 (NA) — Standard deviation was not calculated due to less number of participants. | 10.41 (1.200)

8. Secondary Outcome: Percentage Change From Baseline in Annualized Number of Packed Red Blood Cells (pRBC) Transfusions at Month 24
Description: The annualized number of pRBC transfusions over the 2 year period prior to drug product infusion was compared to the annualized number of pRBC transfusions during the Month 6 to Month 24 period post drug product infusion and the percentage change was reported.
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage of annualized transfusions
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Percentage of annualized transfusions | -100.00 [-100.0 to -20.7] | -65.80 [-96.2 to 2.5] | -90.74 [-100.0 to 2.5]

9. Secondary Outcome: Percentage Change From Baseline in Average Annual Packed Red Blood Cells (pRBC) Transfusion Volume at Month 24
Description: The annualized volume of pRBC transfusions over the 2 year period prior to drug product infusion was compared to the annualized volume of pRBC transfusions in the Month 6 to Month 24 period post drug product Infusion and the percentage change from baseline was reported.
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage of pRBC transfusion volume
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Percentage of pRBC transfusion volume | -100.00 [-100.0 to -26.8] | -71.97 [-97.8 to -8.3] | -92.38 [-100.0 to -8.3]

10. Secondary Outcome: Weighted Average Nadir Hemoglobin (Hb)
Description: Weighted average Hb nadir was defined as an average area under the curve where the Hb closest but within 3 days prior to a transfusion is used as the Hb nadir. If there is a period of more than 60 days without a pRBC transfusion, all Hb records between Day 61 and day of last visit or next transfusion (inclusive) were also considered as nadirs. The weighted average nadir Hb during the period of Month 6 to Month 24 was compared to the weighted average nadir Hb during the 2 years prior to enrollment.
Time Frame: Baseline, Month 6 to Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Grams per deciliter (g/dL)
  Baseline | 8.73 (1.014) | 9.38 (0.431) | 9.02 (0.855)
  Month 6 to Month 24 | 9.97 (1.678) | 8.67 (0.617) | 9.39 (1.446)

11. Secondary Outcome: Number of Participants With Successful Neutrophil Engraftment
Description: Neutrophil engraftment was defined as achieving 3 consecutive absolute neutrophil count (ANC) >= 0.5 × 10^9/L on different days after a post-transplant value of < 0.5 × 10^9/L within 42 days after drug product infusion.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Participants | 10 | 8 | 18

12. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment was defined as the time to the first of 3 consecutive absolute neutrophil count (ANC) >= 0.5 × 10^9/L obtained on different days after a post-transplant value of < 0.5 × 10^9/L. The Day of neutrophil engraftment is the first day of the 3 consecutive measurements, where Day 1 is the day of drug product infusion.
Time Frame: From time of drug product infusion up to 24 months
Population: TP included all participants in the ITT population who underwent LentiGlobin BB305 Drug Product infusion.
Measure: Median (Full Range); unit: Days
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Days | 18.5 [14 to 27] | 19.5 [15 to 30] | 18.5 [14 to 30]

13. Secondary Outcome: Number of Participants With Successful Platelet Engraftment
Description: Platelet engraftment was defined as achieving 3 consecutive platelet values >= 20 × 10^9/L on different days after a post-transplant value of < 20 × 10^9/L, while no platelet transfusions administered for 7 days immediately preceding and during the evaluation period.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Participants | 10 | 8 | 18

14. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment was defined as achieving of first 3 consecutive platelet values >= 20 × 10^9/L obtained on different days after a post-transplant value of < 20 × 10^9/L, while no platelet transfusions administered for 7 days immediately preceding and during the evaluation period. The day of platelet engraftment is the first day of the 3 consecutive measurements, where Day 1 is the day of drug product infusion.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 10 | 8 | 18
Days | 50.5 [19 to 191] | 36.0 [31 to 55] | 39.5 [19 to 191]

15. Secondary Outcome: Transplant-related Mortality
Description: Transplant-related mortality was determined by the investigator (any deaths considered related to the transplant.)
Time Frame: Through 100 and 365 days post-LentiGlobin BB305 Drug Product infusion
Population: ITT population included all participants who initiated any study procedures, beginning with mobilization by G-CSF with or without plerixafor.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 19
Participants | 0

16. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from date of LentiGlobin BB305 Drug Product infusion (Day 1) to date of death. Overall survival was censored at the date of last visit if the participant was still alive. Percentage of participants who survived throughout the study were reported.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Overall
Number analyzed (Participants) | 19
Percentage of participants | 100

17. Secondary Outcome: Percentage of Participants Detected With Replication-competent Lentivirus (RCL)
Description: Blood samples were analyzed for detection of RCL using RCL co-culture assay.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Overall
Number analyzed (Participants) | 18
Percentage of participants | 0

18. Secondary Outcome: Number of Participants With Integration Site Analysis (ISA) With >30% Clonal Contribution
Description: Linear amplification-mediated polymerase chain reaction (LAM-PCR) coupled with next generation sequencing and subsequent (semi-) automated data mining allowed high-throughput analysis of vector integration site (IS) in blood cells from treated participants at multiple time points. ISs detected in peripheral blood cells at early time points generally were due to the expansion of transduced short-term progenitor stem cell clones, and gradually shift to include sites detected due to expansion of transduced long-term stem cell clones. An efficient transduction procedure was anticipated to give rise to a polyclonal population in the participant, reflected by the detection of multiple IS. Additionally, ISA allowed monitoring of the relative contribution of individual clones over time. Number of participants who had IS that contributed to >=30% of the total clones at any time was used as a first step to investigating whether clonal dominance was achieved.
Time Frame: From time of drug product infusion up to 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 18
Participants
  Yes | 0
  No | 18

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE was any AE, occurring at any dose and regardless of causality that: results in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect.
Time Frame: From signing of informed consent to 24 months after the drug product infusion
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Non-β0/β0 | β0/β0 | Overall
Number analyzed (Participants) | 11 | 8 | 19
Participants
  Adverse Events | 10 | 8 | 18
  Serious Adverse Events | 6 | 4 | 10

ADVERSE EVENTS:
Time Frame: From signing of informed consent to 24 months after the drug product infusion
Description: ITT population included all participants who initiated any study procedures, beginning with mobilization by GCSF with or without plerixafor.
Arm/Group | Non-β0/β0 | β0/β0 | Overall
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8 | 0/19
Serious Adverse Events (participants affected / at risk) | 6/11 | 4/8 | 10/19
Other Adverse Events (participants affected / at risk) | 10/11 | 8/8 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-β0/β0 (N=11) | β0/β0 (N=8) | Overall (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 1 | 2
Appendicitis (Infections and infestations) | 1 | 0 | 1
Asymptomatic HIV infection (Infections and infestations) | 1 | 0 | 1
Cat scratch disease (Infections and infestations) | 0 | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-β0/β0 (N=11) | β0/β0 (N=8) | Overall (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 8 | 18
Anaemia (Blood and lymphatic system disorders) | 9 | 8 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 11
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 10
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 6
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 2
Myopia (Eye disorders) | 0 | 1 | 1
Punctate keratitis (Eye disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 8 | 5 | 13
Nausea (Gastrointestinal disorders) | 7 | 5 | 12
Vomiting (Gastrointestinal disorders) | 4 | 7 | 11
Constipation (Gastrointestinal disorders) | 4 | 5 | 9
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 6
Toothache (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Gastritis (Gastrointestinal disorders) | 2 | 0 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 2
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 4 | 5 | 9
Fatigue (General disorders) | 4 | 2 | 6
Pyrexia (General disorders) | 3 | 2 | 5
Non-cardiac chest pain (General disorders) | 2 | 1 | 3
Pain (General disorders) | 1 | 2 | 3
Chest discomfort (General disorders) | 1 | 1 | 2
Catheter site haemorrhage (General disorders) | 1 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 1 | 1
Cyst (General disorders) | 1 | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0 | 1
Dysplasia (General disorders) | 1 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Periportal sinus dilatation (Hepatobiliary disorders) | 0 | 1 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 4
Anal abscess (Infections and infestations) | 1 | 1 | 2
Paronychia (Infections and infestations) | 2 | 0 | 2
Anorectal infection bacterial (Infections and infestations) | 1 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Moraxella infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Syphilis (Infections and infestations) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 6 | 4 | 10
Transfusion reaction (Injury, poisoning and procedural complications) | 6 | 3 | 9
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 2
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Citrate toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 1
Iron overload (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 3
Blood bilirubin increased (Investigations) | 3 | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Blood follicle stimulating hormone increased (Investigations) | 0 | 1 | 1
Blood iron increased (Investigations) | 0 | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 1
Carbon dioxide decreased (Investigations) | 1 | 0 | 1
Forced expiratory flow decreased (Investigations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1
Mean cell haemoglobin concentration increased (Investigations) | 0 | 1 | 1
Mean cell volume decreased (Investigations) | 1 | 0 | 1
Monocyte count decreased (Investigations) | 0 | 1 | 1
Protein total decreased (Investigations) | 0 | 1 | 1
Red blood cell count increased (Investigations) | 1 | 0 | 1
Reticulocyte count decreased (Investigations) | 1 | 0 | 1
Reticulocyte percentage decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 6 | 4 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4 | 6
Dizziness (Nervous system disorders) | 1 | 2 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 4 | 2 | 6
Agitation (Psychiatric disorders) | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 4 | 6
Menstruation irregular (Reproductive system and breast disorders) | 4 | 0 | 4
Ovarian failure (Reproductive system and breast disorders) | 2 | 0 | 2
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 9
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 8 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Palpable purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Sweat gland disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Flushing (Vascular disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT01745120/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT01745120/SAP_001.pdf